CLINICAL TRIAL: NCT02862678
Title: Predictive Value of Diffusion-weighted MRI Performed in Early Post-treatment in the Occurrence of Tumor Recurrence or Progression in Head and Neck Squamous Cell Carcinoma Treated With Chemoradiotherapy: a Pilot Study
Acronym: ORODIFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA13048
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2020-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

ARMS (1):
- Patients with head and neck squamous cell carcinoma (Experimental)
  Interventions: Other: diffusion-weighted MRI

INTERVENTIONS:
Other: diffusion-weighted MRI — Two diffusion-weighted MRI will be performed (one 8 days before chemoradiotherapy treatment and one 3 months after the end of chemoradiotherapy treatment).

SUMMARY:
Head and neck squamous cell carcinoma are frequent. The chemoradiotherapy protocols are part of the reference treatment of locally advanced stage tumors. Diffusion-weighted MRI (DW-MRI) is a non radiating imaging, not requiring injection of gadolinium, giving informations on tumor activity, based on the brownian motion of water molecules. The differences in motion are expressed by the apparent diffusion coefficient (ADC). The ADC variations reflect changes in water molecules motion and redistribution between the intra- and extracellular compartments. Several studies have shown that malignant lesions have an ADC coefficient lowered as compared to benign lesions.

DETAILED DESCRIPTION:
study the diagnostic performance of diffusion MRI performed in early post treatment, notably changes in the ADC factor, in the onset of tumor recurrence or progression in patients showing no residual tumor at the end a treatment by chemoradiotherapy for squamous cell carcinoma of head and neck seat.

compare the characteristics of diffusion MRI, such as ADC coefficient, between patients with residual tumor and patients with no residual tumor after chemoradiotherapy for squamous cell carcinoma of head and neck location.

ELIGIBILITY:
Inclusion Criteria:

* patients with head and neck squamous cell carcinoma
* patients with indication of a treatment by chemoradiotherapy (without surgical indication)
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

* patients with contraindications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-04; Primary Completion 2019-03-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
tumor recurrence | 12 months
  positive histological sample to squamous cell carcinoma between 6 and 12 months after treatment by radiochemotherapy

SECONDARY OUTCOMES:
residual tumors | 6 months
  positive histological sample to squamous cell carcinoma in the 6 months after treatment by radiochemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Background] Brenet E, Barbe C, Hoeffel C, Dubernard X, Merol JC, Fath L, Servagi-Vernat S, Labrousse M. Predictive Value of Early Post-Treatment Diffusion-Weighted MRI for Recurrence or Tumor Progression of Head and Neck Squamous Cell Carcinoma Treated with Chemo-Radiotherapy. Cancers (Basel). 2020 May 14;12(5):1234. doi: 10.3390/cancers12051234. PMID 32422975